CLINICAL TRIAL: NCT02460458
Title: Type 3 Von Willebrand International Registries Inhibitor Prospective Study
Acronym: 3WINTERS-IPS
Status: Completed | Type: Observational
Sponsor: Fondazione Angelo Bianchi Bonomi (Other)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Other Study IDs: ABB-11-01
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Type 3 Von Willebrand's Disease
Keywords: Factor VIII; Hemorrhage; Type 3 Von Willebrand's Disease; Von Willebrand Factor; Von Willebrand's Disease; Hemostasis; Gastro-Intestinal Bleeds
MeSH Terms: conditions — von Willebrand Disease, Type 3; Hemophilia A; Hemorrhage; von Willebrand Diseases | interventions — von Willebrand Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Venous blood sample, that will be used to obtain both citrated Platelet Poor Plasma for Von Willebrand Factor (VWF) assays and Cell Pellet for DNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 3 Von Willebrand's Disease (VWD3): Patients with diagnosis of Type 3 Von Willebrand's Disease
  Interventions: Drug: Von Willebrand Factor

INTERVENTIONS:
Drug: Von Willebrand Factor — Replacement therapy with plasma-derived and/or recombinant VWF concentrates on-demand or under prophylaxis therapeutic scheme.
  Other Names: Plasma-derived and/or recombinantVon Willebrand Factor (VWF) concentrates

SUMMARY:
International Registries and Prospective Study on Type 3 Von Willebrand's Disease (VWD3), aimed to assess number, types and risk factors for bleeding and the efficacy and safety of plasma-derived and/or recombinant Von Willebrand Factor (VWF) concentrates used to treat VWD patients.

DETAILED DESCRIPTION:
Von Willebrand's Disease (VWD) is the most common inherited bleeding disorder, characterized by a quantitative and/or qualitative deficiency of Von Willebrand Factor (VWF), that plays a major role in early phases of hemostasis. Type 3 Von Willebrand's Disease (VWD3) is due to virtually complete deficiency of VWF and, for this reason, has been also described as "severe VWD". Recurrent Gastro-Intestinal Bleeds (GIB) is one of the most challenging complications encountered in the management of patients with VWD. The commonest cause is angiodysplasia (ANGDYS), but often no cause is identified due to the difficulty in making the diagnosis. In recent years, research from several laboratories has identified multiple roles for VWF in the control of vascular function. Globally, these findings provide the first possible explanation for the presence of ANGDYS in patients with VWD. These vascular malformations in the gastrointestinal (GI) tract are characterized by fragile, leaky mucosal vessels. Combined with the hemostatic dysfunction, these can lead to severe intractable bleeding including GIB. VWD3 is inherited as a recessive trait and heterozygous relatives have mild or no bleeding symptoms. Even if the prevalence of VWD3 is very low, the highest rate is found in Iran and the lowest in southern Europe. However, the actual prevalence of VWD3 is still unknown in most countries, due to the lack of retrospective or prospective studies. Although rare, VWD3 is of major interest because of its severe clinical presentation, the need for replacement therapy with plasma-derived and/or recombinant VWF concentrates and the risk of occurrence of anti-VWF inhibitors after the infusion of VWF concentrates, for which risk factors have not been systematically determined.

The major objectives of the study are: to create an international network among European and Iranian Centers (ratio 1:1), the prospective enrollment of at least 250 VWD3 patients using a common database online, the collection of detailed information about previous bleedings and exposure to plasma-derived and/or recombinant VWF concentrates, the use of bleeding severity score of VWD3 calculated with a common questionnaire, the collection of plasma and DNA samples from all the identified VWD3 patients enrolled for centralized analyses, the confirmation of the local VWD3 diagnosis using centralized tests, Evaluation of VWF gene defects, VWF phenotype and risk of anti-VWF inhibitors through common methods, the evaluation of potential correlations between phenotypic results (including markers of angiogenesis) and GIB occurrence, the objective evaluation of severity of GIB in VWD3 patients, the assessment of frequency and sites of bleeding in VWD3 patients followed-up for 2 prospective observation periods (2 years each: 2017-2018 and 2020-2022), the efficacy assessment of the plasma-derived and/or recombinant VWF concentrates used to treat VWD3 (on demand versus prophylaxis) using the most objective criteria for efficacy during 2 prospective observation periods (2 years each: 2017-2018 and 2020-2022), the evaluation of the efficacy and safety of plasma-derived and/or recombinant VWF concentrates in the treatment of GIB during 2 prospective observation periods (2 years each: 2017-2018 and 2020-2022), in comparison to the use of anti-angiogenetic agents within the standard clinical setting.

To these purposes, a cohort of at least 250 patients with diagnosis of VWD3 will be enrolled using homogenous and standardized criteria.

The work planned to achieve the objectives of the project will be divided in three parts:

* the first part deals with standardized criteria for enrolment and collection of retrospective clinical and laboratory data, to be confirmed by centralized laboratories;
* the second part involves a further characterization of clinical and laboratory parameters, collected in the retrospective phase, including prevalence of anti-VWF inhibitors, advanced laboratory tests to further identify VWD3, mutations analyses of the VWF gene;
* the third part of the study is divided in two parts: a first prospective observation and a second prospective observation. The third part for the first time deals with the prospective clinical observation in a large cohort of VWD3 patients all previously well characterized by an international panel of experts.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of any age, including infants, children, adolescent and adults
* Informed Consent obtained (parents should sign for patients < 18 y.o.)
* Previous Diagnosis of VWD3 (VWF Antigen: undetectable or <5 U/dL)
* Detailed information on inherited pattern, history of bleeding, previous exposure to blood products
* Availability of plasma and DNA samples

Exclusion Criteria:

• VWD3 patients who may not be available for follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A large cohort of patients with diagnosis of Type 3 Von Willebrand's Disease (VWD3), enrolled in Europe and in Iran using homogeneous and standardized criteria.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Augusto B. Federici, MD, Study Director — Hematology and Transfusion Medicine, L. Sacco University Hospital, University of Milan, Via G. B. Grassi, 74 20157 Milan, Italy
Locations (25):
- Helsinki University Central Hospital, Department Internal Medicine, Coagulation Disorders, at Haematology and Laboratory Services, Helsinki, Finland
- France (2):
  - Institut d'Hématologie - Hôpital Cardiologique - University of Lille - Haematology Department, Lille
  - Centre Régional de Traitement de l'Hémophilie - Laboratoire d'Hématologie, Nantes
- Germany (3):
  - University Clinic Bonn - Institute of Experimental Haematology & Transfusion Medicine, Bonn
  - University Children's Hospital - Department of Pediatric Hematology and Oncology, Hamburg
  - Department of Haematology, Haemostasis, Oncology and Stem Cell Transplantation - Hannover Medical School - Haemophilia Care Centre, Hanover
- St. Istvan & St. Laszlo Hospital of Budapest - Hematology and Stem Cell Transplantation, Budapest, Hungary
- Iran (7):
  - Ahvaz Jundishpur University of Medical Sciences - Research Center for Thalassemia & Hemoglobinopathy - Division of Hematology & Oncology, Ahvāz
  - Seid-ol-Shohada Hospital - Hemophilia Center - Esfahan University of Medical Science, Isfahan
  - Hemophilia- Thalassaemia Center of Mashhad (Sarvar Clinic) - Mashad University of Medical Science, Mashhad
  - Nemazee Hospital Hemophilia Center - Shiraz University of Medical Science, Shiraz
  - Iranian Hemophilia Comprehensive Treatment Centre - Iranian Hemophilia Society, Tehran
  - Mofid Comprehensive Care Centre for Children with Hemophilia - Shahid Beheshti University of Medical Science, Tehran
  - Thrombosis Hemostasis Research Center - Vali-Asr Hospital - Emam Khmeini Complex Hospital - Tehran University of Medical Science, Tehran
- Italy (5):
  - Azienda Ospedaliera Policlinico Consorziale di Bari - Unità Operativa Semplice di Emostasi e Trombosi, Bari
  - Azienda Ospedaliera Universitaria Careggi - Agenzia per l'Emofilia - Centro di Riferimento Coagulopatie Congenite, Florence
  - Centro Emofilia e Trombosi - Fondazione Angelo Bianchi Bonomi - IRCCS Ospedale Ca' Granda - Dip. di Medicina Interna - Università degli Studi di Milano, Milan
  - Dipartimento di Biotecnologie Cellulari ed Ematologia - Università "Sapienza" di Roma - Policlinico Umberto I, Roma
  - Dipartimento di Terapie Cellulari ed Ematologia - Centro Malattie Emorragiche e Trombotiche - Ospedale San Bortolo, Vicenza
- Netherlands (2):
  - Leiden University Medical Center - Department of Hematology - Hemostasis and Thrombosis Center, Leiden
  - Erasmus Medical Center - Department of Hematology, Rotterdam
- Spain (2):
  - Complejo Hospitalario Universitario de A Coruña - Servicio de Hematología y Hemoterapia, A Coruña
  - Hospital Universitari General Vall d'Hebron - Unidad de Hemofilia, Barcelona
- Lund University - Centre for Thrombosis and Haemostasis - Skane University Hospital, Malmo, Sweden
- Central Manchester University Hospital NHS Foundation Trust - Manchester Royal Infirmary - Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eikenboom JC. Congenital von Willebrand disease type 3: clinical manifestations, pathophysiology and molecular biology. Best Pract Res Clin Haematol. 2001 Jun;14(2):365-79. doi: 10.1053/beha.2001.0139. PMID 11686105
- [Background] Sadler JE, Budde U, Eikenboom JC, Favaloro EJ, Hill FG, Holmberg L, Ingerslev J, Lee CA, Lillicrap D, Mannucci PM, Mazurier C, Meyer D, Nichols WL, Nishino M, Peake IR, Rodeghiero F, Schneppenheim R, Ruggeri ZM, Srivastava A, Montgomery RR, Federici AB; Working Party on von Willebrand Disease Classification. Update on the pathophysiology and classification of von Willebrand disease: a report of the Subcommittee on von Willebrand Factor. J Thromb Haemost. 2006 Oct;4(10):2103-14. doi: 10.1111/j.1538-7836.2006.02146.x. Epub 2006 Aug 2. PMID 16889557
- [Background] Nilsson IM. Commentary to Erik von Willebrand's original paper from 1926 'Hereditar pseudohemofili'. Haemophilia. 1999 May;5(3):220-1. doi: 10.1046/j.1365-2516.1999.0320a.x. No abstract available. PMID 10444292
- [Background] NILSSON IM, BLOMBACK M, BLOMBACK B. v. Willebrand's disease in Sweden; its pathogenesis and treatment. Acta Med Scand. 1959 Jun 30;164:263-78. No abstract available. PMID 14427267
- [Background] Mannucci PM, Bloom AL, Larrieu MJ, Nilsson IM, West RR. Atherosclerosis and von Willebrand factor. I. Prevalence of severe von Willebrand's disease in western Europe and Israel. Br J Haematol. 1984 May;57(1):163-9. doi: 10.1111/j.1365-2141.1984.tb02876.x. PMID 6609712
- [Background] Weiss HJ, Ball AP, Mannucci PM. Incidence of severe von Willebrand's disease. N Engl J Med. 1982 Jul 8;307(2):127. doi: 10.1056/NEJM198207083070222. No abstract available. PMID 6979706
- [Background] Berliner SA, Seligsohn U, Zivelin A, Zwang E, Sofferman G. A relatively high frequency of severe (type III) von Willebrand's disease in Israel. Br J Haematol. 1986 Mar;62(3):535-43. doi: 10.1111/j.1365-2141.1986.tb02966.x. PMID 3082350
- [Background] Iorio A, Oliovecchio E, Morfini M, Mannucci PM; Association of Italian Hemophilia Centres Directors. Italian Registry of Haemophilia and Allied Disorders. Objectives, methodology and data analysis. Haemophilia. 2008 May;14(3):444-53. doi: 10.1111/j.1365-2516.2008.01679.x. Epub 2008 Mar 18. PMID 18355268
- [Background] Federici AB, Mannucci PM. Management of inherited von Willebrand disease in 2007. Ann Med. 2007;39(5):346-58. doi: 10.1080/07853890701513738. PMID 17701477
- [Background] Silwer J. von Willebrand's disease in Sweden. Acta Paediatr Scand Suppl. 1973;238:1-159. No abstract available. PMID 4550005
- [Background] Lak M, Peyvandi F, Mannucci PM. Clinical manifestations and complications of childbirth and replacement therapy in 385 Iranian patients with type 3 von Willebrand disease. Br J Haematol. 2000 Dec;111(4):1236-9. doi: 10.1046/j.1365-2141.2000.02507.x. PMID 11167767
- [Background] Federici AB, Castaman G, Mannucci PM; Italian Association of Hemophilia Centers (AICE). Guidelines for the diagnosis and management of von Willebrand disease in Italy. Haemophilia. 2002 Sep;8(5):607-21. doi: 10.1046/j.1365-2516.2002.00672.x. PMID 12199668
- [Background] Rodeghiero F, Castaman G, Tosetto A, Batlle J, Baudo F, Cappelletti A, Casana P, De Bosch N, Eikenboom JC, Federici AB, Lethagen S, Linari S, Srivastava A. The discriminant power of bleeding history for the diagnosis of type 1 von Willebrand disease: an international, multicenter study. J Thromb Haemost. 2005 Dec;3(12):2619-26. doi: 10.1111/j.1538-7836.2005.01663.x. PMID 16359502
- [Background] Tosetto A, Rodeghiero F, Castaman G, Goodeve A, Federici AB, Batlle J, Meyer D, Fressinaud E, Mazurier C, Goudemand J, Eikenboom J, Schneppenheim R, Budde U, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Lethagen S, Pasi J, Hill F, Peake I. A quantitative analysis of bleeding symptoms in type 1 von Willebrand disease: results from a multicenter European study (MCMDM-1 VWD). J Thromb Haemost. 2006 Apr;4(4):766-73. doi: 10.1111/j.1538-7836.2006.01847.x. PMID 16634745
- [Background] Cattaneo M, Federici AB, Lecchi A, Agati B, Lombardi R, Stabile F, Bucciarelli P. Evaluation of the PFA-100 system in the diagnosis and therapeutic monitoring of patients with von Willebrand disease. Thromb Haemost. 1999 Jul;82(1):35-9. PMID 10456451
- [Background] Mannucci PM, Lattuada A, Castaman G, Lombardi R, Colibretti ML, Ciavarella N, Rodeghiero F. Heterogeneous phenotypes of platelet and plasma von Willebrand factor in obligatory heterozygotes for severe von Willebrand disease. Blood. 1989 Nov 15;74(7):2433-6. PMID 2804373
- [Background] Mannucci PM, Federici AB. Antibodies to von Willebrand factor in von Willebrand disease. Adv Exp Med Biol. 1995;386:87-92. doi: 10.1007/978-1-4613-0331-2_7. No abstract available. PMID 8851017
- [Background] Federici AB. Clinical and molecular markers of inherited von Willebrand disease type 3: are deletions of the VWF gene associated with alloantibodies to VWF? J Thromb Haemost. 2008 Oct;6(10):1726-8. doi: 10.1111/j.1538-7836.2008.03146.x. No abstract available. PMID 18853484
- [Background] Veltkamp JJ, van Tilburg NH. Detection of heterozygotes for recessive von Willebrand's disease by the assay of antihemophilic-factor-like antigen. N Engl J Med. 1973 Oct 25;289(17):882-5. doi: 10.1056/NEJM197310252891703. No abstract available. PMID 4542316
- [Background] Shelton-Inloes BB, Chehab FF, Mannucci PM, Federici AB, Sadler JE. Gene deletions correlate with the development of alloantibodies in von Willebrand disease. J Clin Invest. 1987 May;79(5):1459-65. doi: 10.1172/JCI112974. PMID 3033024
- [Background] Ngo KY, Glotz VT, Koziol JA, Lynch DC, Gitschier J, Ranieri P, Ciavarella N, Ruggeri ZM, Zimmerman TS. Homozygous and heterozygous deletions of the von Willebrand factor gene in patients and carriers of severe von Willebrand disease. Proc Natl Acad Sci U S A. 1988 Apr;85(8):2753-7. doi: 10.1073/pnas.85.8.2753. PMID 3258663
- [Background] Schneppenheim R, Krey S, Bergmann F, Bock D, Budde U, Lange M, Linde R, Mittler U, Meili E, Mertes G, et al. Genetic heterogeneity of severe von Willebrand disease type III in the German population. Hum Genet. 1994 Dec;94(6):640-52. doi: 10.1007/BF00206958. PMID 7989040
- [Background] Eikenboom JC, Castaman G, Vos HL, Bertina RM, Rodeghiero F. Characterization of the genetic defects in recessive type 1 and type 3 von Willebrand disease patients of Italian origin. Thromb Haemost. 1998 Apr;79(4):709-17. PMID 9569178
- [Background] Schneppenheim R, Castaman G, Federici AB, Kreuz W, Marschalek R, Oldenburg J, Oyen F, Budde U. A common 253-kb deletion involving VWF and TMEM16B in German and Italian patients with severe von Willebrand disease type 3. J Thromb Haemost. 2007 Apr;5(4):722-8. doi: 10.1111/j.1538-7836.2007.02460.x. Epub 2007 Feb 26. PMID 17371490
- [Background] Peake IR, Liddell MB, Moodie P, Standen G, Mancuso DJ, Tuley EA, Westfield LA, Sorace JM, Sadler JE, Verweij CL, et al. Severe type III von Willebrand's disease caused by deletion of exon 42 of the von Willebrand factor gene: family studies that identify carriers of the condition and a compound heterozygous individual. Blood. 1990 Feb 1;75(3):654-61. PMID 2297569
- [Background] Mancuso DJ, Tuley EA, Castillo R, de Bosch N, Mannucci PM, Sadler JE. Characterization of partial gene deletions in type III von Willebrand disease with alloantibody inhibitors. Thromb Haemost. 1994 Aug;72(2):180-5. PMID 7831648
- [Background] Baronciani L, Cozzi G, Canciani MT, Peyvandi F, Srivastava A, Federici AB, Mannucci PM. Molecular characterization of a multiethnic group of 21 patients with type 3 von Willebrand disease. Thromb Haemost. 2000 Oct;84(4):536-40. PMID 11057846
- [Background] Mohl A, Marschalek R, Masszi T, Nagy E, Obser T, Oyen F, Sallai K, Bodo I, Schneppenheim R. An Alu-mediated novel large deletion is the most frequent cause of type 3 von Willebrand disease in Hungary. J Thromb Haemost. 2008 Oct;6(10):1729-35. doi: 10.1111/j.1538-7836.2008.03107.x. Epub 2008 Jul 28. PMID 18665926
- [Background] Xie F, Wang X, Cooper DN, Chuzhanova N, Fang Y, Cai X, Wang Z, Wang H. A novel Alu-mediated 61-kb deletion of the von Willebrand factor (VWF) gene whose breakpoints co-locate with putative matrix attachment regions. Blood Cells Mol Dis. 2006 May-Jun;36(3):385-91. doi: 10.1016/j.bcmd.2006.03.003. Epub 2006 May 11. PMID 16690331
- [Background] Cooper DN, Krawczak M. The mutational spectrum of single base-pair substitutions causing human genetic disease: patterns and predictions. Hum Genet. 1990 Jun;85(1):55-74. doi: 10.1007/BF00276326. PMID 2192981
- [Background] Zhang ZP, Lindstedt M, Falk G, Blomback M, Egberg N, Anvret M. Nonsense mutations of the von Willebrand factor gene in patients with von Willebrand disease type III and type I. Am J Hum Genet. 1992 Oct;51(4):850-8. PMID 1415226
- [Background] Eikenboom JC, Ploos van Amstel HK, Reitsma PH, Briet E. Mutations in severe, type III von Willebrand's disease in the Dutch population: candidate missense and nonsense mutations associated with reduced levels of von Willebrand factor messenger RNA. Thromb Haemost. 1992 Oct 5;68(4):448-54. PMID 1448779
- [Background] Bahnak BR, Lavergne JM, Rothschild C, Meyer D. A stop codon in a patient with severe type III von Willebrand disease. Blood. 1991 Aug 15;78(4):1148-9. No abstract available. PMID 1868248
- [Background] Zhang ZP, Falk G, Blomback M, Egberg N, Anvret M. Identification of a new nonsense mutation in the von Willebrand factor gene in patients with von Willebrand disease type III. Hum Mol Genet. 1992 Apr;1(1):61-2. doi: 10.1093/hmg/1.1.61. No abstract available. PMID 1301136
- [Background] Zhang ZP, Blomback M, Egberg N, Falk G, Anvret M. Characterization of the von Willebrand factor gene (VWF) in von Willebrand disease type III patients from 24 families of Swedish and Finnish origin. Genomics. 1994 May 1;21(1):188-93. doi: 10.1006/geno.1994.1241. PMID 8088787
- [Background] Hagiwara T, Inaba H, Yoshida S, Nagaizumi K, Arai M, Hanabusa H, Fukutake K. A novel mutation Gly 1672-->Arg in type 2A and a homozygous mutation in type 2B von Willebrand disease. Thromb Haemost. 1996 Aug;76(2):253-7. PMID 8865541
- [Background] Gupta PK, Saxena R, Adamtziki E, Budde U, Oyen F, Obser T, Schneppenheim R. Genetic defects in von Willebrand disease type 3 in Indian and Greek patients. Blood Cells Mol Dis. 2008 Sep-Oct;41(2):219-22. doi: 10.1016/j.bcmd.2008.03.004. Epub 2008 May 16. PMID 18485763
- [Background] Casana P, Martinez F, Haya S, Lorenzo JI, Espinos C, Aznar JA. Q1311X: a novel nonsense mutation of putative ancient origin in the von Willebrand factor gene. Br J Haematol. 2000 Nov;111(2):552-5. doi: 10.1046/j.1365-2141.2000.02410.x. PMID 11122100
- [Background] Surdhar GK, Enayat MS, Lawson S, Williams MD, Hill FG. Homozygous gene conversion in von Willebrand factor gene as a cause of type 3 von Willebrand disease and predisposition to inhibitor development. Blood. 2001 Jul 1;98(1):248-50. doi: 10.1182/blood.v98.1.248. No abstract available. PMID 11439975
- [Background] Baronciani L, Cozzi G, Canciani MT, Peyvandi F, Srivastava A, Federici AB, Mannucci PM. Molecular defects in type 3 von Willebrand disease: updated results from 40 multiethnic patients. Blood Cells Mol Dis. 2003 May-Jun;30(3):264-70. doi: 10.1016/s1079-9796(03)00033-0. PMID 12737944
- [Background] Gupta PK, Adamtziki E, Budde U, Jaiprakash M, Kumar H, Harbeck-Seu A, Kannan M, Oyen F, Obser T, Wedekind I, Saxena R, Schneppenheim R. Gene conversions are a common cause of von Willebrand disease. Br J Haematol. 2005 Sep;130(5):752-8. doi: 10.1111/j.1365-2141.2005.05660.x. PMID 16115133
- [Background] Eikenboom JC, Vink T, Briet E, Sixma JJ, Reitsma PH. Multiple substitutions in the von Willebrand factor gene that mimic the pseudogene sequence. Proc Natl Acad Sci U S A. 1994 Mar 15;91(6):2221-4. doi: 10.1073/pnas.91.6.2221. PMID 8134377
- [Background] Zhang ZP, Falk G, Blomback M, Egberg N, Anvret M. A single cytosine deletion in exon 18 of the von Willebrand factor gene is the most common mutation in Swedish vWD type III patients. Hum Mol Genet. 1992 Dec;1(9):767-8. doi: 10.1093/hmg/1.9.767. No abstract available. PMID 1302613
- [Background] Xie F, Wang X, Cooper DN, Lan F, Fang Y, Cai X, Wang Z, Wang H. Compound heterozygosity for two novel mutations (1203insG/Y1456X) in the von Willebrand factor gene causing type 3 von Willebrand disease. Haemophilia. 2007 Sep;13(5):645-8. doi: 10.1111/j.1365-2516.2007.01514.x. PMID 17880457
- [Background] Wetzstein V, Budde U, Oyen F, Ding X, Herrmann J, Liebig B, Schneppenheim R. Intracranial hemorrhage in a term newborn with severe von Willebrand disease type 3 associated with sinus venous thrombosis. Haematologica. 2006 Dec;91(12 Suppl):ECR60. PMID 17194666
- [Background] Krawczak M, Cooper DN. Gene deletions causing human genetic disease: mechanisms of mutagenesis and the role of the local DNA sequence environment. Hum Genet. 1991 Mar;86(5):425-41. doi: 10.1007/BF00194629. PMID 2016084
- [Background] Efstratiadis A, Posakony JW, Maniatis T, Lawn RM, O'Connell C, Spritz RA, DeRiel JK, Forget BG, Weissman SM, Slightom JL, Blechl AE, Smithies O, Baralle FE, Shoulders CC, Proudfoot NJ. The structure and evolution of the human beta-globin gene family. Cell. 1980 Oct;21(3):653-68. doi: 10.1016/0092-8674(80)90429-8. PMID 6985477
- [Background] Zhang ZP, Blomback M, Nyman D, Anvret M. Mutations of von Willebrand factor gene in families with von Willebrand disease in the Aland Islands. Proc Natl Acad Sci U S A. 1993 Sep 1;90(17):7937-40. doi: 10.1073/pnas.90.17.7937. PMID 8367445
- [Background] Mohlke KL, Nichols WC, Rehemtulla A, Kaufman RJ, Fagerstrom HM, Ritvanen KL, Kekomaki R, Ginsburg D. A common frameshift mutation in von Willebrand factor does not alter mRNA stability but interferes with normal propeptide processing. Br J Haematol. 1996 Oct;95(1):184-91. doi: 10.1046/j.1365-2141.1996.7572377.x. PMID 8857958
- [Background] Eikenboom JC, Reitsma PH, van der Velden PA, Briet E. Instability of repeats of the von Willebrand factor gene variable number tandem repeat sequence in intron 40. Br J Haematol. 1993 Jul;84(3):533-5. doi: 10.1111/j.1365-2141.1993.tb03114.x. PMID 8105872
- [Background] Antonarakis SE. Recommendations for a nomenclature system for human gene mutations. Nomenclature Working Group. Hum Mutat. 1998;11(1):1-3. doi: 10.1002/(SICI)1098-1004(1998)11:13.0.CO;2-O. No abstract available. PMID 9450896
- [Background] Mertes G, Ludwig M, Finkelnburg B, Krawczak M, Schwaab R, Brackmann HH, Olek K. A G+3-to-T donor splice site mutation leads to skipping of exon 50 in von Willebrand factor mRNA. Genomics. 1994 Nov 1;24(1):190-1. doi: 10.1006/geno.1994.1602. No abstract available. PMID 7896280
- [Background] Zhang Z, Lindstedt M, Blomback M, Anvret M. Effects of the mutant von Willebrand factor gene in von Willebrand disease. Hum Genet. 1995 Oct;96(4):388-94. doi: 10.1007/BF00191794. PMID 7557958
- [Background] Allen S, Abuzenadah AM, Hinks J, Blagg JL, Gursel T, Ingerslev J, Goodeve AC, Peake IR, Daly ME. A novel von Willebrand disease-causing mutation (Arg273Trp) in the von Willebrand factor propeptide that results in defective multimerization and secretion. Blood. 2000 Jul 15;96(2):560-8. PMID 10887119
- [Background] Castaman G, Lattuada A, Mannucci PM, Rodeghiero F. Factor VIII:C increases after desmopressin in a subgroup of patients with autosomal recessive severe von Willebrand disease. Br J Haematol. 1995 Jan;89(1):147-51. doi: 10.1111/j.1365-2141.1995.tb08921.x. PMID 7833254
- [Background] Tjernberg P, Castaman G, Vos HL, Bertina RM, Eikenboom JC. Homozygous C2362F von Willebrand factor induces intracellular retention of mutant von Willebrand factor resulting in autosomal recessive severe von Willebrand disease. Br J Haematol. 2006 May;133(4):409-18. doi: 10.1111/j.1365-2141.2006.06055.x. PMID 16643449
- [Background] Castaman G, Eikenboom JC, Lattuada A, Mannucci PM, Rodeghiero F. Heightened proteolysis of the von Willebrand factor subunit in patients with von Willebrand disease hemizygous or homozygous for the C2362F mutation. Br J Haematol. 2000 Jan;108(1):188-90. doi: 10.1046/j.1365-2141.2000.01807.x. PMID 10651743
- [Background] Baronciani L, Federici AB, Cozzi G, La Marca S, Punzo M, Rubini V, Canciani MT, Mannucci PM. Expression studies of missense mutations p.D141Y, p.C275S located in the propeptide of von Willebrand factor in patients with type 3 von Willebrand disease. Haemophilia. 2008 May;14(3):549-55. doi: 10.1111/j.1365-2516.2008.01682.x. Epub 2008 Mar 4. PMID 18328061
- [Background] Voorberg J, Fontijn R, Calafat J, Janssen H, van Mourik JA, Pannekoek H. Assembly and routing of von Willebrand factor variants: the requirements for disulfide-linked dimerization reside within the carboxy-terminal 151 amino acids. J Cell Biol. 1991 Apr;113(1):195-205. doi: 10.1083/jcb.113.1.195. PMID 2007623
- [Background] Peake IR, Bowen D, Bignell P, Liddell MB, Sadler JE, Standen G, Bloom AL. Family studies and prenatal diagnosis in severe von Willebrand disease by polymerase chain reaction amplification of a variable number tandem repeat region of the von Willebrand factor gene. Blood. 1990 Aug 1;76(3):555-61. PMID 2378985
- [Background] Federici AB, Mazurier C, Berntorp E, Lee CA, Scharrer I, Goudemand J, Lethagen S, Nitu I, Ludwig G, Hilbert L, Mannucci PM. Biologic response to desmopressin in patients with severe type 1 and type 2 von Willebrand disease: results of a multicenter European study. Blood. 2004 Mar 15;103(6):2032-8. doi: 10.1182/blood-2003-06-2072. Epub 2003 Nov 20. PMID 14630825
- [Background] Castaman G, Lethagen S, Federici AB, Tosetto A, Goodeve A, Budde U, Batlle J, Meyer D, Mazurier C, Fressinaud E, Goudemand J, Eikenboom J, Schneppenheim R, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Pasi J, Hill F, Peake I, Rodeghiero F. Response to desmopressin is influenced by the genotype and phenotype in type 1 von Willebrand disease (VWD): results from the European Study MCMDM-1VWD. Blood. 2008 Apr 1;111(7):3531-9. doi: 10.1182/blood-2007-08-109231. Epub 2008 Jan 29. PMID 18230755
- [Background] Cattaneo M, Moia M, Delle Valle P, Castellana P, Mannucci PM. DDAVP shortens the prolonged bleeding times of patients with severe von Willebrand disease treated with cryoprecipitate. Evidence for a mechanism of action independent of released von Willebrand factor. Blood. 1989 Nov 1;74(6):1972-5. PMID 2508791
- [Background] Mannucci PM, Chediak J, Hanna W, Byrnes J, Ledford M, Ewenstein BM, Retzios AD, Kapelan BA, Schwartz RS, Kessler C; Alphanate Study Group. Treatment of von Willebrand disease with a high-purity factor VIII/von Willebrand factor concentrate: a prospective, multicenter study. Blood. 2002 Jan 15;99(2):450-6. doi: 10.1182/blood.v99.2.450. PMID 11781224
- [Background] Federici AB, Baudo F, Caracciolo C, Mancuso G, Mazzucconi MG, Musso R, Schinco PC, Targhetta R, Mannuccio Mannucci P. Clinical efficacy of highly purified, doubly virus-inactivated factor VIII/von Willebrand factor concentrate (Fanhdi) in the treatment of von Willebrand disease: a retrospective clinical study. Haemophilia. 2002 Nov;8(6):761-7. doi: 10.1046/j.1365-2516.2002.00688.x. PMID 12410644
- [Background] Bello IF, Yuste VJ, Molina MQ, Navarro FH. Fanhdi, efficacy and safety in von Willebrand's disease: prospective international study results. Haemophilia. 2007 Dec;13 Suppl 5:25-32. doi: 10.1111/j.1365-2516.2007.01570.x. PMID 18078394
- [Background] Federici AB, Barillari G, Zanon E, Mazzucconi MG, Musso R, Targhetta R, Mannucci PM. Efficacy and safety of highly purified, doubly virus-inactivated VWF/FVIII concentrates in inherited von Willebrand's disease: results of an Italian cohort study on 120 patients characterized by bleeding severity score. Haemophilia. 2010 Jan;16(1):101-10. doi: 10.1111/j.1365-2516.2009.02088.x. Epub 2009 Oct 6. PMID 19811543
- [Background] Dobrkovska A, Krzensk U, Chediak JR. Pharmacokinetics, efficacy and safety of Humate-P in von Willebrand disease. Haemophilia. 1998;4 Suppl 3:33-9. doi: 10.1046/j.1365-2516.1998.0040s3033.x. PMID 10028316
- [Background] Lillicrap D, Poon MC, Walker I, Xie F, Schwartz BA; Association of Hemophilia Clinic Directors of Canada. Efficacy and safety of the factor VIII/von Willebrand factor concentrate, haemate-P/humate-P: ristocetin cofactor unit dosing in patients with von Willebrand disease. Thromb Haemost. 2002 Feb;87(2):224-30. PMID 11858481
- [Background] Franchini M, Rossetti G, Tagliaferri A, Pattacini C, Pozzoli D, Lippi G, Manzato F, Bertuzzo D, Gandini G. Efficacy and safety of factor VIII/von Willebrand's factor concentrate (Haemate-P) in preventing bleeding during surgery or invasive procedures in patients with von Willebrand disease. Haematologica. 2003 Nov;88(11):1279-83. PMID 14607757
- [Background] Federici AB, Castaman G, Franchini M, Morfini M, Zanon E, Coppola A, Tagliaferri A, Boeri E, Mazzucconi MG, Rossetti G, Mannucci PM. Clinical use of Haemate P in inherited von Willebrand's disease: a cohort study on 100 Italian patients. Haematologica. 2007 Jul;92(7):944-51. doi: 10.3324/haematol.11124. PMID 17606445
- [Background] Gill JC, Ewenstein BM, Thompson AR, Mueller-Velten G, Schwartz BA; Humate-P Study Group. Successful treatment of urgent bleeding in von Willebrand disease with factor VIII/VWF concentrate (Humate-P): use of the ristocetin cofactor assay (VWF:RCo) to measure potency and to guide therapy. Haemophilia. 2003 Nov;9(6):688-95. doi: 10.1046/j.1351-8216.2003.00816.x. PMID 14750934
- [Background] Thompson AR, Gill JC, Ewenstein BM, Mueller-Velten G, Schwartz BA; Humate-P Study Group. Successful treatment for patients with von Willebrand disease undergoing urgent surgery using factor VIII/VWF concentrate (Humate-P). Haemophilia. 2004 Jan;10(1):42-51. doi: 10.1046/j.1351-8216.2003.00809.x. PMID 14962219
- [Background] Lethagen S, Kyrle PA, Castaman G, Haertel S, Mannucci PM; HAEMATE P Surgical Study Group. von Willebrand factor/factor VIII concentrate (Haemate P) dosing based on pharmacokinetics: a prospective multicenter trial in elective surgery. J Thromb Haemost. 2007 Jul;5(7):1420-30. doi: 10.1111/j.1538-7836.2007.02588.x. Epub 2007 Apr 16. PMID 17439628
- [Background] Stadler M, Gruber G, Kannicht C, Biesert L, Radomski KU, Suhartono H, Pock K, Neisser-Svae A, Weinberger J, Romisch J, Svae TE. Characterisation of a novel high-purity, double virus inactivated von Willebrand Factor and Factor VIII concentrate (Wilate). Biologicals. 2006 Dec;34(4):281-8. doi: 10.1016/j.biologicals.2005.11.010. Epub 2006 Feb 23. PMID 16500114
- [Background] Favaloro EJ, Lloyd J, Rowell J, Baker R, Rickard K, Kershaw G, Street A, Scarff K, Barrese G, Maher D, McLachlan AJ. Comparison of the pharmacokinetics of two von Willebrand factor concentrates [Biostate and AHF (High Purity)] in people with von Willebrand disorder. A randomised cross-over, multi-centre study. Thromb Haemost. 2007 Jun;97(6):922-30. PMID 17549293
- [Background] Shortt J, Dunkley S, Rickard K, Baker R, Street A. Efficacy and safety of a high purity, double virus inactivated factor VIII/von Willebrand factor concentrate (Biostate) in patients with von Willebrand disorder requiring invasive or surgical procedures. Haemophilia. 2007 Mar;13(2):144-8. doi: 10.1111/j.1365-2516.2006.01430.x. PMID 17286766
- [Background] Menache D, Aronson DL, Darr F, Montgomery RR, Gill JC, Kessler CM, Lusher JM, Phatak PD, Shapiro AD, Thompson AR, White GC 2nd. Pharmacokinetics of von Willebrand factor and factor VIIIC in patients with severe von Willebrand disease (type 3 VWD): estimation of the rate of factor VIIIC synthesis. Cooperative Study Groups. Br J Haematol. 1996 Sep;94(4):740-5. doi: 10.1046/j.1365-2141.1996.d01-1860.x. PMID 8826903
- [Background] Goudemand J, Scharrer I, Berntorp E, Lee CA, Borel-Derlon A, Stieltjes N, Caron C, Scherrmann JM, Bridey F, Tellier Z, Federici AB, Mannucci PM. Pharmacokinetic studies on Wilfactin, a von Willebrand factor concentrate with a low factor VIII content treated with three virus-inactivation/removal methods. J Thromb Haemost. 2005 Oct;3(10):2219-27. doi: 10.1111/j.1538-7836.2005.01435.x. PMID 16194199
- [Background] Borel-Derlon A, Federici AB, Roussel-Robert V, Goudemand J, Lee CA, Scharrer I, Rothschild C, Berntorp E, Henriet C, Tellier Z, Bridey F, Mannucci PM. Treatment of severe von Willebrand disease with a high-purity von Willebrand factor concentrate (Wilfactin): a prospective study of 50 patients. J Thromb Haemost. 2007 Jun;5(6):1115-24. doi: 10.1111/j.1538-7836.2007.02562.x. PMID 17403090
- [Background] Bergamaschini L, Mannucci PM, Federici AB, Coppola R, Guzzoni S, Agostoni A. Posttransfusion anaphylactic reactions in a patient with severe von Willebrand disease: role of complement and alloantibodies to von Willebrand factor. J Lab Clin Med. 1995 Mar;125(3):348-55. PMID 7897302
- [Background] Ciavarella N, Schiavoni M, Valenzano E, Mangini F, Inchingolo F. Use of recombinant factor VIIa (NovoSeven) in the treatment of two patients with type III von Willebrand's disease and an inhibitor against von Willebrand factor. Haemostasis. 1996;26 Suppl 1:150-4. doi: 10.1159/000217258. PMID 8904191
- [Background] Boyer-Neumann C, Dreyfus M, Wolf M, Veyradier A, Meyer D. Multi-therapeutic approach to manage delivery in an alloimmunized patient with type 3 von Willebrand disease. J Thromb Haemost. 2003 Jan;1(1):190-2. doi: 10.1046/j.1538-7836.2003.00009.x. No abstract available. PMID 12871560
- [Background] Berntorp E, Petrini P. Long-term prophylaxis in von Willebrand disease. Blood Coagul Fibrinolysis. 2005 Apr;16 Suppl 1:S23-6. doi: 10.1097/01.mbc.0000167659.23262.18. PMID 15849523
- [Background] De Meyer SF, Vanhoorelbeke K, Chuah MK, Pareyn I, Gillijns V, Hebbel RP, Collen D, Deckmyn H, VandenDriessche T. Phenotypic correction of von Willebrand disease type 3 blood-derived endothelial cells with lentiviral vectors expressing von Willebrand factor. Blood. 2006 Jun 15;107(12):4728-36. doi: 10.1182/blood-2005-09-3605. Epub 2006 Feb 14. PMID 16478886
- [Background] von Willebrand EA. (1926) Hereditär Pseudohemofili. Finska Läkaresällskapets Handlingar 68, 87-112.
- [Background] Federici AB, Bucciarelli P, Castaman G et al. (2007) Incidence and determinants of bleeding in different types of von Willebrand disease:results of the first prospective multicenter study on 814 Italian patients Blood 110, 713
- [Background] Abuzenadah AM, Gursel T, Ingerslev J et al. (1999) Mutational analysis of the von Willebrand factor gene in 27 families from Turkey with von Willebrand disease Thromb Haemost 82 (Suppl), 283
- [Background] Castaman G, Giacomelli SH, Coppola A et al. (2008) Molecular bases of type 3 von Willebrand disease in Italy: report on 12 families Blood Transfus Suppl 3, 44
- [Background] Gazda H, Budde U, Krey S et al. (1997) Delta C in exon 18 of the von Willebrand factor gene is the most common mutation in patients with severe von Willebrand disease type 3 in Poland Blood 90 (Suppl 1), 94b
- [Background] Titapiwatanakun R, Guenther JC, Asmann YW et al. (2007) Novel Mutations in Types 2 & 3 von Willebrand Disease and Correlation with von Willebrand Factor Multimer Patterns. Blood 110, 2136
- [Background] Montgomery RR, Jozwiak MA, Hutter JJ et al. (1999) A homozygous variant of the von Willebrand factor (VWF) that fails to c-terminal dimerize resulting in loss of VWF multimers larger than dimer Blood 94 (Suppl 1), 443a
- [Background] Schneppenheim R, Budde U, Drewke E et al. (1999) Cysteine mutations of von Willebrand factor correlate with different types of von Willebrand disease Thromb Haemost 82 (Suppl), 283
- [Background] Enayat MS, Guilliatt AM, Surdhar GK et al. (2001) Identification of five novel mutations in families with type 3 von Willebrand's disease Thromb Haemost 86 (Suppl), P1810
- [Background] Mannucci PM. Treatment of von Willebrand's Disease. N Engl J Med. 2004 Aug 12;351(7):683-94. doi: 10.1056/NEJMra040403. No abstract available. PMID 15306670
- [Background] Federici AB, Gianniello F, Canciani MT et al. (2005) Secondary long-term prophylaxis in severe patients with von Willebrand disease: an Italian cohort study Blood 106, 507a
- [Background] Marchese M, De Cristofaro R, Federici AB, Biondi A, Petruzziello L, Tringali A, Spada C, Mutignani M, Ronconi P, Costamagna G. Duodenal and gastric Dieulafoy's lesions in a patient with type 2A von Willebrand's disease. Gastrointest Endosc. 2005 Feb;61(2):322-5. doi: 10.1016/s0016-5107(04)02636-7. No abstract available. PMID 15729257
- [Background] Tosetto A, Rodeghiero F, Castaman G, Bernardi M, Bertoncello K, Goodeve A, Federici AB, Batlle J, Meyer D, Mazurier C, Goudemand J, Eikenboom J, Schneppenheim R, Budde U, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Lethagen S, Pasi J, Hill F, Peake I. Impact of plasma von Willebrand factor levels in the diagnosis of type 1 von Willebrand disease: results from a multicenter European study (MCMDM-1VWD). J Thromb Haemost. 2007 Apr;5(4):715-21. doi: 10.1111/j.1538-7836.2007.02444.x. PMID 17408405
- [Background] Federici AB. Highly purified VWF/FVIII concentrates in the treatment and prophylaxis of von Willebrand disease: the PRO. WILL Study. Haemophilia. 2007 Dec;13 Suppl 5:15-24. doi: 10.1111/j.1365-2516.2007.01573.x. PMID 18078393
- [Background] Federici AB, Mannucci PM, Castaman G, Baronciani L, Bucciarelli P, Canciani MT, Pecci A, Lenting PJ, De Groot PG. Clinical and molecular predictors of thrombocytopenia and risk of bleeding in patients with von Willebrand disease type 2B: a cohort study of 67 patients. Blood. 2009 Jan 15;113(3):526-34. doi: 10.1182/blood-2008-04-152280. Epub 2008 Sep 19. PMID 18805962
- [Background] Gritti G, Cortelezzi A, Bucciarelli P, Rezzonico F, Lonati S, La Marca S, Silvestris I, Federici AB. Circulating and progenitor endothelial cells are abnormal in patients with different types of von Willebrand disease and correlate with markers of angiogenesis. Am J Hematol. 2011 Aug;86(8):650-6. doi: 10.1002/ajh.22070. Epub 2011 May 31. PMID 21630316
- [Background] Abshire TC, Federici AB, Alvarez MT, Bowen J, Carcao MD, Cox Gill J, Key NS, Kouides PA, Kurnik K, Lail AE, Leebeek FW, Makris M, Mannucci PM, Winikoff R, Berntorp E; VWD PN. Prophylaxis in severe forms of von Willebrand's disease: results from the von Willebrand Disease Prophylaxis Network (VWD PN). Haemophilia. 2013 Jan;19(1):76-81. doi: 10.1111/j.1365-2516.2012.02916.x. Epub 2012 Jul 23. PMID 22823000
- [Background] Castaman G, Goodeve A, Eikenboom J; European Group on von Willebrand Disease. Principles of care for the diagnosis and treatment of von Willebrand disease. Haematologica. 2013 May;98(5):667-74. doi: 10.3324/haematol.2012.077263. PMID 23633542
- [Background] Federici AB, Bucciarelli P, Castaman G, Mazzucconi MG, Morfini M, Rocino A, Schiavoni M, Peyvandi F, Rodeghiero F, Mannucci PM. The bleeding score predicts clinical outcomes and replacement therapy in adults with von Willebrand disease. Blood. 2014 Jun 26;123(26):4037-44. doi: 10.1182/blood-2014-02-557264. Epub 2014 Apr 30. PMID 24786773
- [Background] Abdul-Kadir R, McLintock C, Ducloy AS, El-Refaey H, England A, Federici AB, Grotegut CA, Halimeh S, Herman JH, Hofer S, James AH, Kouides PA, Paidas MJ, Peyvandi F, Winikoff R. Evaluation and management of postpartum hemorrhage: consensus from an international expert panel. Transfusion. 2014 Jul;54(7):1756-68. doi: 10.1111/trf.12550. Epub 2014 Mar 12. PMID 24617726
- [Background] Makris M, Federici AB, Mannucci PM, Bolton-Maggs PHB, Yee TT, Abshire T, Berntorp E. The natural history of occult or angiodysplastic gastrointestinal bleeding in von Willebrand disease. Haemophilia. 2015 May;21(3):338-342. doi: 10.1111/hae.12571. Epub 2014 Nov 7. PMID 25381842
- [Background] Federici AB. Clinical and laboratory diagnosis of VWD. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):524-30. doi: 10.1182/asheducation-2014.1.524. Epub 2014 Nov 18. PMID 25696905
- [Background] Holm E, Abshire TC, Bowen J, Alvarez MT, Bolton-Maggs P, Carcao M, Federici AB, Gill JC, Halimeh S, Kempton C, Key NS, Kouides P, Lail A, Landorph A, Leebeek F, Makris M, Mannucci P, Mauser-Bunschoten EP, Nugent D, Valentino LA, Winikoff R, Berntorp E. Changes in bleeding patterns in von Willebrand disease after institution of long-term replacement therapy: results from the von Willebrand Disease Prophylaxis Network. Blood Coagul Fibrinolysis. 2015 Jun;26(4):383-8. doi: 10.1097/MBC.0000000000000257. PMID 25688461
- [Background] Randi AM, Laffan MA. Von Willebrand factor and angiogenesis: basic and applied issues. J Thromb Haemost. 2017 Jan;15(1):13-20. doi: 10.1111/jth.13551. PMID 27778439
- [Background] Federici AB. Current and emerging approaches for assessing von Willebrand disease in 2016. Int J Lab Hematol. 2016 May;38 Suppl 1:41-9. doi: 10.1111/ijlh.12540. PMID 27426859
- [Background] De Jong A, Eikenboom J. Developments in the diagnostic procedures for von Willebrand disease. J Thromb Haemost. 2016 Mar;14(3):449-60. doi: 10.1111/jth.13243. Epub 2016 Feb 12. PMID 26714181
- [Background] Abshire T, Cox-Gill J, Kempton CL, Leebeek FW, Carcao M, Kouides P, Donfield S, Berntorp E. Prophylaxis escalation in severe von Willebrand disease: a prospective study from the von Willebrand Disease Prophylaxis Network. J Thromb Haemost. 2015 Sep;13(9):1585-9. doi: 10.1111/jth.12995. Epub 2015 Jul 14. PMID 25930155
- [Background] Engelen ET, van Galen KP, Schutgens RE. Thalidomide for treatment of gastrointestinal bleedings due to angiodysplasia: a case report in acquired von Willebrand syndrome and review of the literature. Haemophilia. 2015 Jul;21(4):419-29. doi: 10.1111/hae.12701. Epub 2015 Apr 30. PMID 25929157
- [Background] Franchini M, Mannucci PM. Gastrointestinal angiodysplasia and bleeding in von Willebrand disease. Thromb Haemost. 2014 Sep 2;112(3):427-31. doi: 10.1160/TH13-11-0952. Epub 2014 Jun 5. PMID 24898873
- [Background] Randi AM, Laffan MA, Starke RD. Von Willebrand factor, angiodysplasia and angiogenesis. Mediterr J Hematol Infect Dis. 2013 Sep 2;5(1):e2013060. doi: 10.4084/MJHID.2013.060. PMID 24106610
- [Background] Thachil J, Hay CR, Campbell S. Tamoxifen for recurrent bleeds due to angiodysplasia in von Willebrand's disease. Haemophilia. 2013 Sep;19(5):e313-5. doi: 10.1111/hae.12196. Epub 2013 Jun 4. No abstract available. PMID 23731407
- [Background] Castaman G, Federici AB, Tosetto A, La Marca S, Stufano F, Mannucci PM, Rodeghiero F. Different bleeding risk in type 2A and 2M von Willebrand disease: a 2-year prospective study in 107 patients. J Thromb Haemost. 2012 Apr;10(4):632-8. doi: 10.1111/j.1538-7836.2012.04661.x. PMID 22329792
- [Background] Starke RD, Ferraro F, Paschalaki KE, Dryden NH, McKinnon TA, Sutton RE, Payne EM, Haskard DO, Hughes AD, Cutler DF, Laffan MA, Randi AM. Endothelial von Willebrand factor regulates angiogenesis. Blood. 2011 Jan 20;117(3):1071-80. doi: 10.1182/blood-2010-01-264507. Epub 2010 Nov 3. PMID 21048155
- [Background] Veyradier A, Balian A, Wolf M, Giraud V, Montembault S, Obert B, Dagher I, Chaput JC, Meyer D, Naveau S. Abnormal von Willebrand factor in bleeding angiodysplasias of the digestive tract. Gastroenterology. 2001 Feb;120(2):346-53. doi: 10.1053/gast.2001.21204. PMID 11159874
- [Background] Bowers M, McNulty O, Mayne E. Octreotide in the treatment of gastrointestinal bleeding caused by angiodysplasia in two patients with von Willebrand's disease. Br J Haematol. 2000 Mar;108(3):524-7. doi: 10.1046/j.1365-2141.2000.01897.x. PMID 10759709
- [Background] Van Belle E, Rauch A, Vincent F, Robin E, Kibler M, Labreuche J, Jeanpierre E, Levade M, Hurt C, Rousse N, Dally JB, Debry N, Dallongeville J, Vincentelli A, Delhaye C, Auffray JL, Juthier F, Schurtz G, Lemesle G, Caspar T, Morel O, Dumonteil N, Duhamel A, Paris C, Dupont-Prado A, Legendre P, Mouquet F, Marchant B, Hermoire S, Corseaux D, Moussa K, Manchuelle A, Bauchart JJ, Loobuyck V, Caron C, Zawadzki C, Leroy F, Bodart JC, Staels B, Goudemand J, Lenting PJ, Susen S. Von Willebrand Factor Multimers during Transcatheter Aortic-Valve Replacement. N Engl J Med. 2016 Jul 28;375(4):335-44. doi: 10.1056/NEJMoa1505643. PMID 27464202
- [Background] Susen S, Rauch A, Van Belle E, Vincentelli A, Lenting PJ. Circulatory support devices: fundamental aspects and clinical management of bleeding and thrombosis. J Thromb Haemost. 2015 Oct;13(10):1757-67. doi: 10.1111/jth.13120. Epub 2015 Sep 25. PMID 26302994
- [Background] Blatchford O, Murray WR, Blatchford M. A risk score to predict need for treatment for upper-gastrointestinal haemorrhage. Lancet. 2000 Oct 14;356(9238):1318-21. doi: 10.1016/S0140-6736(00)02816-6. PMID 11073021
- [Background] Gerson LB, Fidler JL, Cave DR, Leighton JA. ACG Clinical Guideline: Diagnosis and Management of Small Bowel Bleeding. Am J Gastroenterol. 2015 Sep;110(9):1265-87; quiz 1288. doi: 10.1038/ajg.2015.246. Epub 2015 Aug 25. PMID 26303132
- [Background] Strate LL, Gralnek IM. ACG Clinical Guideline: Management of Patients With Acute Lower Gastrointestinal Bleeding. Am J Gastroenterol. 2016 Apr;111(4):459-74. doi: 10.1038/ajg.2016.41. Epub 2016 Mar 1. PMID 26925883
- [Background] Jackson CS, Gerson LB. Management of gastrointestinal angiodysplastic lesions (GIADs): a systematic review and meta-analysis. Am J Gastroenterol. 2014 Apr;109(4):474-83; quiz 484. doi: 10.1038/ajg.2014.19. Epub 2014 Mar 18. PMID 24642577
- [Background] Martin-Grace J, Tamagno G. Somatostatin analogs in the medical management of occult bleeding of the lower digestive tract. Gastroenterol Res Pract. 2015;2015:702921. doi: 10.1155/2015/702921. Epub 2015 Mar 9. PMID 25838821
- [Background] Holleran G, Hall B, Breslin N, McNamara D. Long-acting somatostatin analogues provide significant beneficial effect in patients with refractory small bowel angiodysplasia: Results from a proof of concept open label mono-centre trial. United European Gastroenterol J. 2016 Feb;4(1):70-6. doi: 10.1177/2050640614559121. Epub 2015 Nov 5. PMID 26966525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2012 - March 2015
Groups:
- Type 3 Von Willebrand's Disease (VWD3): Patients with diagnosis of Type 3 Von Willebrand's Disease (VWD3). In the Retrospective Phase, the retrospective data of the participants were collected and analyzed, and a blood sample was drawn. During the Confirmatory Phase, local VWD3 diagnosis was verified using centralized tests. Participants with a confirmed case of VWD3 were then prospectively observed for two years (First Prospective Phase). After a Confirmation of the Clinical Phase Data, the participants started a Second Prospective Phase, being observed for two additional years.
Period: Retrospective Phase
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Started | 265
Completed | 265
Not Completed | 0
Period: Confirmatory Phase
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Started | 265
Completed | 210
Not Completed | 55
Not completed — Patients excluded basing on phenotype central analysis | 31
Not completed — Lack of sample to analyse | 19
Not completed — Patients excluded due to lack of central characterized VWD mutations | 5
Period: First Prospective Phase
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Started | 210
Completed | 126
Not Completed | 84
Not completed — Lost to Follow-up | 84
Period: Confirmation of Clinical Phase Data
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Started | 126
Completed | 92
Not Completed | 34
Not completed — Lost to Follow-up | 34

BASELINE CHARACTERISTICS:
Population: The study population includes a cohort of 265 patients with local diagnosis of Type 3 Von Willebrand's Disease (VWD3) enrolled using homogeneous and standardized criteria.
Groups:
- Type 3 Von Willebrand's Disease (VWD3): Patients with diagnosis of Type 3 Von Willebrand's Disease (VWD3)
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75
  Between 18 and 65 years | 179
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.19 (18.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 9
  Sweden | 3
  Hungary | 16
  Finland | 9
  Italy | 60
  United Kingdom | 8
  France | 13
  Germany | 18
  Iran, Islamic Republic of | 119
  Spain | 10
MCMDM-1 Bleeding Score System Retrospective Data [Mean (Full Range); unit: units on a scale] — Range from -1 to +4 for each symptom considered (12 symptoms, total range from -12 to 48). For each symptom: 0=no symptom, 1=referred by the patient, 2=brought to medical attention, 3=major intervention. Score 0 and 1 are attributed to symptoms referred by the patient, hence without any precise medical intervention. Population: The MCMDM-1 Bleeding Score System Retrospective Data was collected for 249 / 265 patients since historical data about bleedings was not fully available at the investigational sites for the remaining 16 patients.
  units on a scale
    number analyzed (Participants) | 249
    (all) | 15.14 [1 to 48]

OUTCOME MEASURES:

1. Primary Outcome: Centralized Factor VIII (FVIII) Procoagulant Activity (FVIII:C) Laboratory Test for Type 3 Von Willebrand's Disease (VWD3) Diagnosis
Description: Measurement of the Factor VIII (FVIII) Procoagulant Activity (FVIII:C) in the blood through one-stage clotting test. Only patients with FVIII:C less or equal to 5 IU/dL were considered for the analysis.
Time Frame: 12 months (confirmatory phase)
Population: Factor VIII (FVIII) Procoagulant Activity (FVIII:C) was centrally obtained from samples collected from investigational sites.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 183
IU/dL | 2.42 (0.88)

2. Primary Outcome: Centralized Von Willebrand Factor Antigen (VWF:Ag) Laboratory Test for Type 3 Von Willebrand's Disease (VWD3) Diagnosis
Description: Measurement of the amount of Von Willebrand Factor (VWF) protein in the blood through Von Willebrand Factor Antigen (VWF:Ag) test. Only patients with VWF:Ag less or equal to 5 IU/dL were considered for the analysis.
Time Frame: 12 months (confirmatory phase)
Population: Von Willebrand Factor (VWF) protein blood levels were centrally obtained from samples collected from investigational sites.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 209
IU/dL | 1.01 (1.03)

3. Primary Outcome: Centralized Factor VIII (FVIII) Amidolytic Activity (FVIII:Am) Laboratory Test for Type 3 Von Willebrand's Disease (VWD3) Diagnosis
Description: Measurement of Factor VIII (FVIII) Amidolytic Activity (FVIII:Am) in the blood through chromogenic test. Only patients with FVIII:Am less or equal to 5 IU/dL were considered for the analysis.
Time Frame: 12 months (confirmatory phase)
Population: Factor VIII (FVIII) Amidolytic Activity (FVIII:Am) in the blood was centrally obtained from samples collected from investigational sites.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 191
IU/dL | 1.54 (0.91)

4. Primary Outcome: Centralized Factor VIII (FVIII) Antigen (FVIII:Ag) Laboratory Test for Type 3 Von Willebrand's Disease (VWD3) Diagnosis
Description: Measurement of the amount of Factor VIII (FVIII) protein in the blood through FVIII:Ag test. Only patients with FVIII:Ag less or equal to 5 IU/dL were considered for the analysis.
Time Frame: 12 months (confirmatory phase)
Population: Factor VIII (FVIII) protein blood levels were centrally obtained from samples collected from investigational sites.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 140
IU/dL | 3.63 (0.83)

5. Primary Outcome: Centralized Von Willebrand Factor (VWF) Multimer Analysis for Type 3 Von Willebrand's Disease (VWD3) Diagnosis
Description: Multimer analysis of Von Willebrand Factor (VWF) was carried out by electrophoresis of blood samples collected by investigational sites. The number of patients belonging of each multimer profile group (1 - Homozygotes / 2 - Only Protomers / 3 - 2-4 Bands) was calculated. The qualitative evaluation of VWF multimers is part of the diagnostic process of VWD3.
Time Frame: 12 months (confirmatory phase)
Population: Von Willebrand Factor (VWF) multimer profiles of patients were centrally obtained from samples collected from investigational sites.
Measure: Count of Participants; unit: Participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 243
Participants
  Homozygotes | 174
  Only Protomers | 15
  2 - 4 Bands | 54

6. Primary Outcome: Centralized Von Willebrand Factor (VWF) Propeptide Laboratory Test for Type 3 Von Willebrand's Disease (VWD3) Diagnosis
Description: Measurement of Von Willebrand Factor (VWF) Propeptide levels in the blood through VWF Propeptide test. This test has been performed according to the most recent methods and the results are important to characterize the molecular aspects of VWD patients.
Time Frame: 12 months (confirmatory phase)
Population: Von Willebrand Factor (VWF) Propeptide blood levels were centrally obtained from samples collected from investigational sites.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 238
IU/dL | 6.44 (13.98)

7. Primary Outcome: Centralized Molecular Type 3 Von Willebrand's Disease (VWD3) Diagnosis Through DNA Analysis
Description: Evaluation of the presence of Von Willebrand Factor (VWF) gene defects (confirmation or screening for the first time).
Time Frame: 12 months (confirmatory phase)
Population: Samples were not available for 34 patients out of 265
Measure: Count of Participants; unit: Participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 231
Participants
  Analyzed participants with confirmed VWD3 diagnosis | 219
  Analyzed participants without confirmed VWD3 diagnosis | 12

8. Primary Outcome: Record of Bleeding Episodes
Description: Record of all bleedings occurred during the prospective phase of the study.
Time Frame: 24 months (first prospective phase) + 24 months (second prospective phase)
Population: Patients that have competed both prospective phases.
Measure: Number; unit: bleeding episodes
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 92
bleeding episodes | 713

9. Primary Outcome: Adverse Events
Description: Record of all adverse events occurred during the prospective phase of the study.
Time Frame: 24 months (first prospective phase) + 24 months (second prospective phase)
Population: Patients that have competed both prospective phases.
Measure: Number; unit: AE
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 92
AE | 47

10. Primary Outcome: Type of Von Willebrand Factor / Factor VIII (VWF/FVIII)-Containing Concentrates in Use
Description: Record of any Von Willebrand Factor / Factor VIII (VWF/FVIII)-containing concentrates used and currently in use, including the current schedule type of treatment.
Time Frame: 24 months (first prospective phase) + 24 months (second prospective phase)
Population: Patients that have competed both prospective phases.
Measure: Number; unit: participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 92
participants
  Recombinant Activated Factor FVIII | 1
  Fanhdi | 1
  Voncento/Haemate P | 33
  Wilate/Wilfactin (Wilfact) | 5
  Aryoseven | 1

11. Secondary Outcome: Patients Experiencing Allergic Reactions During Use of Von Willebrand Factor (VWF)-Containing Concentrates
Description: Record of any allergic and anaphylactic reactions occurred in the past due to the use of any Von Willebrand Factor (VWF) concentrate and the date of onset.
Time Frame: 24 months (retrospective phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 265
Participants | 41

12. Secondary Outcome: Number of Participants With Previous Use of Blood Products
Description: Record of any product used during the retrospective phase (collected type of blood products/Von Willebrand Factor (VWF) concentrate, year of first exposure, units used).
Time Frame: 24 months (retrospective phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 265
Participants
  Packed red cells | 24
  Cryoprecipitates | 123
  Fresh frozen plasma | 10
  Platelet concentrates | 1

13. Secondary Outcome: Number of Patients With Available Local Laboratory Test for Anti-Von Willebrand Factor (Anti-VWF) Antibodies
Description: Evaluation of the titre of Anti-Von Willebrand Factor (anti-VWF) Antibodies through Bethesda Test.
Time Frame: 24 months (retrospective phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 265
Participants | 4

14. Secondary Outcome: Local Laboratory Tests for Type 3 Von Willebrand's Disease (VWD3) Diagnosis (Composite)
Description: Number of patients for who the following tests have been performed:
  Hemoglobin (mmol/L), Hemagglutination Titer (HT) (%), Mean Corpuscular Volume (MVC) (fl), Leucocytes (E9/L), Neutrophils (%), Basophils (%), Eosinophils (%), Lymphocytes (%), Platelet Count (E9/L), Mean Platelet Volume (MPV) (fl), Prothrombin Time (sec), Partial Thromboplastin Time (PTT) (sec), Partial Thromboplastin Time Mix 50:50 (PTT mix 50:50) (sec), Ferritin (ug/l), Bleeding Time (min:sec), Closure Time (sec), Collagen/ADP (sec), Collagen/Epinephrine (sec); Factor VIII Procoagulant Activity (FVIII:C) (IU/mL), Von Willebrand Factor Ristocetin Cofactor (VWF:RCo) (IU/mL), Won Willebrand Factor Antigen (VWF:Ag) (IU/mL).
Time Frame: 24 months (retrospective phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
Number analyzed (Participants) | 265
Participants | 265

ADVERSE EVENTS:
Time Frame: Data about adverse events occurring to participants will be collected throughout the whole study period (retrospective phase + prospective phase).
Description: For adverse events associated with treatments, Investigators are encouraged to contact the manufacturer / regulatory authorities to report it, and to share a copy of any form submitted with Sponsor. An Independent Data Monitoring Committee (DMC) will be appointed for data monitoring on safety.
Arm/Group | Type 3 Von Willebrand's Disease (VWD3)
All-Cause Mortality (participants affected / at risk) | 0/265
Serious Adverse Events (participants affected / at risk) | 5/265
Other Adverse Events (participants affected / at risk) | 28/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 3 Von Willebrand's Disease (VWD3) (N=265)
Post-partum bleeding in uterus (Reproductive system and breast disorders) | 1 (1)
Gastro-Intestinal bleeding (Gastrointestinal disorders) | 1 (1)
Intracranial bleeding (Nervous system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Headache righr hemisphere (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 3 Von Willebrand's Disease (VWD3) (N=265)
Abdomen and flank pain (General disorders) | 1 (1)
Abdominal pain (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 10 (23)
Allergy (Immune system disorders) | 1 (4)
Rhinorrea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthrosis in right ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle trauma (Musculoskeletal and connective tissue disorders) | 1 (1)
B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot burn (Skin and subcutaneous tissue disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Capsulitis in finger (right hand) (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (General disorders) | 2 (2)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 3 (3)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Hypogastric pain (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2)
Pharingitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pelvic pain (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Trauma of elbow (Injury, poisoning and procedural complications) | 1 (1)
Trauma of gum (Injury, poisoning and procedural complications) | 1 (1)
Twisting ankle (Injury, poisoning and procedural complications) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flashing after receiving VWD Concentrate (General disorders) | 1 (1)
In Vitro Fertilization (Reproductive system and breast disorders) | 1 (1)
Sensitiveness (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Lack of data due to issues with samples. Some samples were not collected properly or properly stored, resulting impossible to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT02460458/Prot_SAP_000.pdf